CLINICAL TRIAL: NCT06717906
Title: Comparing Three Modalities (Trans Abdominal, Trans-perineal and Endoscopic Ultrasound) of Ultrasonography for Rectal Imaging in Ulcerative Colitis: The TRINITY Study
Brief Title: Comparing TRIple Rectal Ultrasound Imaging Technology in Ulcerative Colitis
Acronym: TRINITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: AGPL/TRINITY/01; Version:01
Record Dates: First submitted 2024-08-18; First posted 2024-12-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Endosonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patients with Ulcerative colitis (Other): Adult patients (18-75 years) with Ulcerative colitis Pregnant, lactating and acute severe colitis excluded
  Interventions: Diagnostic Test: Endoscopic Ultrasound

INTERVENTIONS:
Diagnostic Test: Endoscopic Ultrasound — If sigmoidoscopy is warranted as per clinical indication, the consenting patients shall undergo endoscopic ultrasound (EUS) using a radial echo-endoscope during the same sitting of sigmoidoscopy without incurring any additional cost to the patient. Total rectal wall thickness in anterior and posterior wall shall be measured in upper, middle and lower rectum with assessment of vascularity (Modified Limberg scale). The maximal wall thickness including maximum mucosal and submucosal thickness shall be noted and compared to total wall thickness measured by transabdominal ultrasound (TAS) and Transperineal ultrasound (TPUS). On sigmoidoscopy, rectal inflammation shall be measured by ulcerative colitis endoscopic index of severity (UCEIS) in rectum. Biopsy seal be taken as standard protocol to document histologic inflammation (measured by Nancy histologic index) which is known to predict future risk of relapse.

SUMMARY:
This study aims to evaluate the correlation of rectal wall thickness and vascularity measurements using trans-abdominal ultrasound (TAS), trans-perineal ultrasound (TPUS), and endoscopic ultrasound (EUS) in adult patients with ulcerative colitis (UC). The primary objective is to correlate rectal total wall thickness measured by TPUS with EUS, while secondary objectives include correlating rectal wall thickness and vascularity as measured by TAS, TPUS, and EUS, with endoscopic and histologic activity. Additionally, the study will assess changes in patient management following EUS/sigmoidoscopy compared to TAS/TPUS alone. Consecutive UC patients attending an IBD clinic will undergo clinical assessment using the Simple Clinical Colitis Activity Index (SCCAI) followed by TAS and TPUS as point-of-care tests. If clinically indicated, patients will also undergo sigmoidoscopy and EUS during the same visit, with measurements compared and correlated to histologic inflammation and fecal calprotectin (FCP) levels when available. This cross-sectional study will include a follow-up period until biopsy results are obtained, with a recruitment duration of 6-12 months and a target sample size of 170 patients (60 patients with mid-end ultrasound machine, rest with high-end ultrasound machine for transabdominal and transperineal ultrasound).

DETAILED DESCRIPTION:
This study is designed to assess the correlation of rectal wall thickness and vascularity measurements obtained through trans-abdominal ultrasound (TAS), trans-perineal ultrasound (TPUS), and endoscopic ultrasound (EUS) in adult patients with ulcerative colitis (UC). The primary goal is to determine how well rectal total wall thickness measured via TPUS correlates with EUS findings. Secondary objectives include comparing rectal wall thickness and vascularity measured by TAS, TPUS, and EUS with endoscopic activity, histologic activity, and fecal calprotectin (FCP) levels. Additionally, the study aims to evaluate changes in patient management resulting from additional investigations, such as sigmoidoscopy and EUS, over the standard TAS and TPUS procedures. UC patients attending an inflammatory bowel disease (IBD) clinic will undergo a clinical assessment using the Simple Clinical Colitis Activity Index (SCCAI), followed by baseline TAS and TPUS, both performed as point-of-care tests. If deemed clinically necessary, patients will also undergo sigmoidoscopy and EUS during the same visit, with rectal wall thickness and vascularity measured across different rectal sections and correlated with histologic inflammation assessed via biopsy and measured by the Nancy histologic index. The study will also explore correlations with FCP levels where data are available. This cross-sectional study includes a follow-up period until biopsy results are obtained, with an estimated recruitment duration of 6-12 months and a target sample size of 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years) with Ulcerative colitis

Exclusion Criteria:

* Pregnant
* Lactating mother
* Endoscopy not required
* No consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Compare diagnostic accuracy of endoscopic ultrasound in predicting endoscopic remission | Baseline
  Wall thickness (in mm) measured by endoscopic ultrasound in predicting endoscopic remission in rectum in ulcerative colitis

SECONDARY OUTCOMES:
Compare diagnostic accuracy of endoscopic ultrasound in predicting histologic remission | Baseline
  Wall thickness (in mm) measured by endoscopic ultrasound in predicting histologic remission in rectum in ulcerative colitis
Compare diagnostic accuracy of endoscopic ultrasound vascularity in predicting histologic remission | Baseline
  Vascularity grades (modified Limberg scale: score 0-3, higher score indicates worse outcome) measured by endoscopic ultrasound in predicting histologic remission in ulcerative colitis
Compare diagnostic accuracy of transperineal ultrasound vascularity in predicting histologic remission | Baseline
  Vascularity grades (modified Limberg score: 0-3, higher score indicates worse outcome) measured by transperineal ultrasound in predicting histologic remission in ulcerative colitis
Compare diagnostic accuracy of transperineal ultrasound in predicting endoscopic remission | Baseline
  Wall thickness (in mm) measured by transperineal ultrasound in predicting endoscopic remission in rectum in ulcerative colitis
Compare diagnostic accuracy of transperineal ultrasound in predicting histlogic remission | Baseline
  Wall thickness (in mm) measured by endoscopic ultrasound in predicting histologic remission in rectum in ulcerative colitis
Compare diagnostic accuracy of endoscopic ultrasound vascularity in predicting endoscopic remission | Baseline
  Vascularity grades (modified Limberg score: 0-3, higher score indicates worse outcome) measured by endoscopic ultrasound in predicting endoscopic remission in rectum in ulcerative colitis
Compare diagnostic accuracy of transperineal ultrasound vascularity in predicting endoscopic remission | Baseline
  Vascularity grades (modified Limberg score: 0-3, higher score indicates worse outcome) measured by transperineal ultrasound in predicting endoscopioc remission in ulcerative colitis

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, India

IPD SHARING:
Plan to Share IPD: No